CLINICAL TRIAL: NCT04042857
Title: Safety and Efficacy of Next Science Wound Gel in the Treatment of Mild to Moderate Distal Subungual Onychomycosis (DSO): An Open-Label Pilot Study
Brief Title: Safety and Efficacy of Next Science Gel on Toenail Fungus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Science TM (Industry)
Collaborators: Doctors Research Network (Unknown); Tissue Analytics (Unknown); NTS Ventures (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-010
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Onychomycosis of Toenail
Keywords: DSO; toenail; onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Next Science (Experimental): Patients will apply Next Science treatment to the study target hallux nail for 48 weeks daily.
  Interventions: Device: Next Science Treatment Gel

INTERVENTIONS:
Device: Next Science Treatment Gel — Next Science Treatment Gel will be applied after nail surface nail-filing and/or debridement.

SUMMARY:
This is a 52 week, 20-patient open-label pilot study on the safety and efficacy of Next Science Wound gel in the treatment of mild to moderate Distal Subungual Onychomycosis.

DETAILED DESCRIPTION:
Patients will apply Next Science Wound Gel daily to each study treatment hallux nail for 48 weeks once approved for participation. Analysis will be attained via potassium hydroxide examination (KOH test), nail culture, PCR analysis, and photographic imaging. Subjects may have both hallux nails sampled at screening for culture and KOH testing if both hallux nails appear to meet the criteria for study inclusion. Only subjects with both a positive culture and KOH examination will start study treatment. Subjects may have repeat KOH and culture testing both performed if the first screening test results in at least one of the tests being negative. At investigator's discretion, other affected toenails besides the study target hallux nail may be treated but will not be included for analysis. Patients will come for in-clinic visits at screening, baseline/randomization visit/week 0, week 4, week 8, week 12, week 24, week 36, week 48, and week 52.

If subjects achieve complete cure (as defined by mycological cure and 0% nail involvement) prior to Week 48, patients will be encouraged to continue in the trial with active treatment for the full protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years old and above
2. Established and active diagnosis of distal subungual onychomycosis of at least one hallux nail affecting 20-75% of the hallux nail
3. Positive culture for dermatophytes and positive potassium hydroxide examination
4. Provide signed and dated informed consent
5. Willing to comply with all study procedures and available for the duration of the study

Exclusion Criteria:

1. Known allergic reaction to the study products
2. Unable to provide signed and dated informed consent form
3. Unable or unwilling to comply with all study procedures and/or unavailable for duration of the study
4. Thickness of mycotic nail is greater than 3mm
5. Less than 2mm of clear nail at the proximal aspect
6. History of rheumatoid arthritis
7. Subject with any other disease or condition other than DSO that would affect nail appearance or interfere with image analysis
8. Unwilling or unable to limit use of nail polish for duration of study
9. Known history of PVD, immune system concerns, or ongoing chemotherapy
10. Severe moccasin tinea pedis
11. Prior systemic antifungal drugs 6 months before study start date
12. Prior topical therapy for toenail fungus 2 months before study start date
13. Any diseases or circumstances in which the patient should not participate in the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Mycological Cure at 48 Weeks | Baseline to 48 Weeks
  Mycological cure rate at week 48 as defined by negative potassium hydroxide examination and negative culture of the target hallux nail
Clinical Efficacy at 48 Weeks | Baseline to 48 Weeks
  Clinical efficacy rate at week 48 as defined by less than 10% clinical involvement of the target hallux nail

SECONDARY OUTCOMES:
Complete Cure at Week 48 | Baseline to 48 Weeks
  Complete cure rate at week 48 defined as 0% clinical involvement, negative potassium hydroxide examination and negative culture of the target hallux nail
Complete Cure at Week 52 | Baseline to 52 Weeks
  Complete cure rate at week 52 defined as 0% clinical involvement, negative mycology, and negative potassium hydroxide examination of the target hallux nail at week 52
Almost Complete Cure at Week 48 | Baseline to 48 Weeks
  Almost complete cure rate at week 48 defined as less than 10% clinical involvement, negative potassium hydroxide examination, and negative culture of the target hallux nail at week 48
Almost Complete Cure at Week 52 | Baseline to Week 52
  Almost complete cure rate at week 52 defined as less than 10% clinical involvement, negative potassium hydroxide examination, and negative culture of the target hallux nail at Week 52
Time to Complete Cure | Baseline to 52 Weeks
  Measured across all observation points
Time to Almost Complete Cure | Baseline to 52 Weeks
  Measured across all observation points
Percent Change in Area of Nail Involvement | Baseline to 52 Weeks
  Calculated as a ratio of clear to involved measured across all observation points
Growth of Clear Nail | Baseline to 52 Weeks
  Change in area of clear nail growth measured across all observation points
Mycological Cure Rate | Baseline to 52 Weeks
  Changes in mycological cure rates (Changes in the proportion of subjects who achieved mycological cure, defined as negative culture and potassium hydroxide examination) measured across all observation points
Dermatopyhyte Identification and Characterization | Baseline to 52 Weeks
  Changes in the types of dermatophytes dermatophytes across all observation points
Overall Fungal Species | Baseline to 52 Weeks
  Change types of overall fungal species across all observation points

CONTACTS AND LOCATIONS:
Overall Officials: Maria S Surprenant, DPM, Principal Investigator — Doctors Research Network
Locations (1):
- Doctors Research Network, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No